CLINICAL TRIAL: NCT00991848
Title: Effect of Intravenous Lidocaine on Manifestations of Fibromyalgia
Brief Title: Lidocaine on Manifestations of Fibromyalgia
Acronym: LIMAFIBRO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Roberto Vlainich, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAF09; NSA
Record Dates: First submitted 2009-10-06; First posted 2009-10-08 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Fibromyalgia; Chronic Pain
Keywords: Lidocaine;; Fibromyalgia; signs; symptoms
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lidocaine (Experimental): Patients received 240 mg lidocaine diluted in 125 mL 0.9% saline. The solutions were infused over a period of 1 h, once a week, for 4 weeks (T1, T2, T3 and T4).
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — received 240 mg lidocaine diluted in 125 mL 0.9% saline.

SUMMARY:
Background and Objectives: Fibromyalgia is a pain syndrome characterized by numerous manifestations. The objective of this study was to evaluate the effect of the combination of intravenous lidocaine and amitriptyline on the manifestations of fibromyalgia. Methods: A prospective, randomized, double-blind, comparative study was conducted. All patient received 25 mg amitriptyline. Patients of group 1 (n = 15) received 125 mL 0.9% saline, and patients of group 2 (n = 15) received 240 mg lidocaine in 125 mL 0.9% saline once a week for 4 weeks. Manifestations were recorded before and 4 weeks after treatment. Pain intensity was rated on a verbal numerical scale.

DETAILED DESCRIPTION:
Amitriptyline was chosen in the present study because it is the most widely used antidepressant with proven analgesic efficacy for the treatment of a variety of chronic pain syndromes. Amitriptyline also promotes improvement of sleep, an effect observed in the present study.

Lidocaine has been widely applied by the intravenous route and patients with a variety of pain syndromes, including fibromyalgia, have reported pain relief with this technique.The dose of lidocaine employed by various investigators ranges from 1 to 5 mg/kg administered over a period of 30-60 min. The minimum effective dose is 1.5 mL/L, which is achieved with 2-5 mg/kg infused over 30-60 min. In these study, 240 mg lidocaine was administered, corresponding to about 3 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* pain in the four quadrants of the body for at least 3 months
* sleep disorders
* fatigue
* subjective edema
* depression
* paresthesia.

Exclusion Criteria:

* alterations in thyroid
* rheumatological
* renal and hepatic function
* trauma
* rheumatic, neuromuscular or psychiatric disease
* infectious arthropathy
* other pain syndromes
* drug hypersensitivity
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2005-01; Primary Completion 2007-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
effect of the combination of intravenous lidocaine and amitriptyline on the clinical manifestations of fibromyalgia | 4 weeks

SECONDARY OUTCOMES:
Pain intensity by numerical scale (0 - 10)where 0 being an absent of pain and 10 measuring as the highest for pain intensity | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rioko K Sakata, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil